CLINICAL TRIAL: NCT00538408
Title: Whole Body Magnetic Resonance Angiography in Patients With Symptomatic Peripheral Ischemia
Brief Title: Whole Body Magnetic Resonance Angiography in Ischemic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Yousef Nielsen, Herlev University Hospital
Other Study IDs: H-D-2007-0041
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Atherosclerosis; Intermittent Claudication
Keywords: Magnetic resonance; whole body; angiography; vasovist; gadofosveset; dotarem; blood pool agent
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication | interventions — gadoterate meglumine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Whole body magnetic resonance angiography (dotarem)
Device: Whole body magnetic resonance angiography (vasovist)

SUMMARY:
To investigate the diagnostic performance of whole body magnetic resonance angiography (WB-MRA) using two different magnetic resonance contrast agents.

DETAILED DESCRIPTION:
Atherosclerosis of the lower leg arteries is a common disease. Patients with this condition has symptoms of ischemia, for instance intermittent claudication (pain during exercise). Diagnosis of atherosclerosis in the legs is normally done with an interventional x-ray-based angiography (DSA- digital subtraction angiography). This is uncomfortable for the patient, and associated with risks of complications (bleeding, vascular damage, embolism).A novel approach to diagnosing atherosclerosis is the use of magnetic resonance angiography. A variant of this is the whole body magnetic resonance angiography(WB-MRA), that produce a picture of the arteries in almost the whole body (excluding the coronary arteries). WB-MRA has a number of advantages compared to DSA. It does not use ionizing radiation, is not invasive, uses a contrast medium with fewer side affects and finally gives a covers a great deal of the arteries in the body.

This study will compare WB-MRA with DSA in patients with symptoms of peripheral atherosclerosis in the lower legs. We will investigate 2 different contrast agents used for WB-MRA. The patients will be randomized to receive either the contrast medium Dotarem or the contrast medium Vasovist. In both groups we will compare the results of WB-MRA with DSA.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity ischemia (claudication, ischemic wounds)
* Referred to digital subtraction angiography (DSA)

Exclusion Criteria:

* Renal insufficiency (GFR < 30 ml/min)
* Contra-indications for MRI-examination (claustrophobia, metal-implants, pacemaker)
* Dementia
* Pregnancy/lactation
* Allergy to gadolinium based MRI contrast agents
* Acute disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Vascular diagnostic quality on the WB-MRA. Degree of arterial stenosis on the WB-MRA.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S Thomsen, Prof., Study Chair — University Hospital at Herlev Copenhagen Denmark
Locations (1):
- Department of Radiology, Herlev University Hospital, Herlev, Copenhagen, Denmark